CLINICAL TRIAL: NCT05480306
Title: Randomized Phase 2 Study of DKN-01 Plus FOLFIRI/FOLFOX and Bevacizumab Versus FOLFIRI/FOLFOX and Bevacizumab as Second-line Treatment of Advanced Colorectal Cancer (DeFianCe)
Brief Title: Phase 2 Study of DKN-01 in Colorectal Cancer
Acronym: DeFianCe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leap Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEK-DKK1-P207
Record Dates: First submitted 2022-07-21; First posted 2022-07-29 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Colorectal Adenocarcinoma; Colo-rectal Cancer; Colorectal Cancer Metastatic
Keywords: DKK1; colorectal cancer; DKN-01
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — IFL protocol; Bevacizumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): DKN-01 + FOLFIRI or FOLFOX + bevacizumab
  Interventions: Drug: DKN-01; Drug: FOLFIRI; Drug: Bevacizumab; Drug: FOLFOX
- Control (Active Comparator): FOLFIRI or FOLFOX + bevacizumab
  Interventions: Drug: FOLFIRI; Drug: Bevacizumab; Drug: FOLFOX

INTERVENTIONS:
Drug: DKN-01 — 30 minute IV infusion (400mg) every two weeks with an additional loading dose in the first cycle of treatment
  Other Names: LY2812176
  Arms: Treatment
Drug: FOLFIRI — 90-min IV infusion of irinotecan, leucovorin, and fluorouracil followed by a continuous 46-hour infusion of fluorouracil every two weeks
Drug: Bevacizumab — 90-min IV infusion (5mg)
Drug: FOLFOX — 2 hour IV infusion of oxaliplatin, folinic acid, and fluorouracil followed by a continuous 46-hour infusion of fluorouracil every two weeks

SUMMARY:
This is a Phase 2 randomized, open-label, two-part, multicenter study with a safety run-in to evaluate efficacy and safety of DKN-01 plus FOLFIRI/FOLFOX and bevacizumab versus standard of care (SOC) [FOLFIRI/FOLFOX and bevacizumab] as second-line treatment of advanced CRC patients.

DETAILED DESCRIPTION:
This is a Phase 2 randomized, open-label, two-part, multicenter study with a safety run-in to evaluate efficacy and safety of DKN-01 plus FOLFIRI/FOLFOX and bevacizumab versus standard of care (SOC) [FOLFIRI/FOLFOX and bevacizumab] as second-line treatment of advanced CRC patients.

In Parts A and B, approximately 200 evaluable adult advanced CRC patients with measurable disease (RECIST v1.1) who have radiographically progressed during or following 1 line of systemic treatment will be enrolled in the study.

The study consists of a Screening Period, a Treatment Period, a Safety Follow-up Period (SFUP) and a Long-Term Follow-up Period (LTFU). Patients will be followed in the SFUP for approximately 30 days (+7 days) after the last administration of study drug and then enter the LTFU period to be followed for survival and subsequent therapies. Additionally, patients that ended study treatment for a reason unrelated to progressive disease [PD] will also be followed for disease progression in the LTFU period.

ELIGIBILITY:
Adult patients with advanced CRC with measurable disease (RECIST v1.1) who have radiographically progressed during or following one line of systemic treatment will be enrolled in the study.

Inclusion Criteria:

Patients meeting all of the following criteria will be considered eligible for study entry:

1. Disease progression following first-line systemic therapy with any fluoropyrimidine-based regimen for advanced disease (except FOLFOXIRI, see exclusion criteria).

   • Patients may have received prior neoadjuvant or adjuvant therapy which could have included irinotecan or oxaliplatin. If progression has occurred within 12 months from last dose of neoadjuvant or adjuvant treatment, this regimen will be considered as the one line of systemic therapy for advanced disease.
   * If assigned to receive FOLFIRI, patient may have received no prior irinotecan as part of first-line systemic therapy.
   * If assigned to receive FOLFOX, patient may have received no prior oxaliplatin as part of first line systemic therapy.
   * Prior treatment with an anti-VEGF or anti-EGFR therapy is allowed as first-line and/or maintenance systemic therapy.
2. Able to provide written informed consent for any study specific procedures.
3. One or more tumors measurable on radiographic imaging as defined by RECIST 1.1
4. Sufficient tumor tissue for mandatory pre-treatment evaluation (fresh biopsy [preferred], or archived tissue block specimen).
5. ECOG performance status ≤1 within 7 days of first dose of study drug. Acceptable liver, renal, hematologic, and coagulation function
6. Females of childbearing potential and male partners of female patients must agree to use adequate contraception during the study and for 6 months after their last dose of study drug

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for study entry:

1. Diagnosis of Microsatellite instability-high (MSI-H)/mismatch repair-deficient (dMMR) and/or BRAF V600E mutation positive colorectal cancer.
2. Prior therapy with an anti-DKK1, FOLFOXIRI, PD-1, anti-PD-L1, anti-PD-L-2 or any other antibody or drug specifically targeting T-cell co-stimulation or coinhibitory checkpoint.
3. Systemic anti-cancer therapy within 28 days prior to first dose of study drug.
4. Major surgery within 28 days prior to first dose of study drug.
5. Prior radiation therapy within 14 days prior to first dose of study drug.
6. Active leptomeningeal disease or uncontrolled brain metastases.
7. Any active cancer ≤ 2 years before first dose of study drug with the exception of cancer for this study.
8. New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, or unstable arrhythmia.
9. Fridericia-corrected QT interval (QTcF) > 470 msec (female) or history of congenital long QT syndrome.
10. Active, uncontrolled bacterial, viral, or fungal infections, within 14 days of study entry requiring systemic therapy.
11. Serious nonmalignant disease
12. Pregnant or nursing.
13. History of osteonecrosis of the hip or have evidence of structural bone abnormalities in the proximal femur on MRI scan that are symptomatic and clinically significant.
14. Known osteoblastic bony metastasis.
15. Major surgery 28 days prior to study entry.
16. Prior radiation therapy within 14 days prior to study entry.
17. Significant allergy to a pharmaceutical therapy that, in the opinion of the Investigator, poses an increased risk to the patient.
18. Active substance abuse.
19. Known dihydropyrimidine dehydrogenase deficiency.
20. Administration of a live vaccine within 28 days before first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | approximately 6 months
  PFS, as determined by the Investigator per RECIST v1.1 of DKN-01 plus SOC versus SOC.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | approximately 6 months
  ORR, as determined by the Investigator per RECIST v1.1 of DKN-01 plus SOC versus SOC
Duration of Response (DoR) | approximately 6 months
  DoR, as determined by the Investigator per RECIST v1.1 of DKN-01 plus SOC versus SOC
Overall Survival (OS) | approximately 6 months
  OS with DKN-01 plus SOC versus SOC
Incidence of ≥Grade 3 related treatment-related adverse events (TRAEs). | approximately 6 months

OTHER OUTCOMES:
Duration of Complete Response (DoCR) | approximately 6 months
  DoCR using RECIST v1.1
Duration of clinical benefit (DoCB) | approximately 6 months
  DoCB as determined using RECIST v1.1, is defined as the time from the date of randomization (or date of registration for Part A patients) to the time of progressive disease or death due to any cause in patients who had a best overall response of complete response (CR), partial response (PR), or stable disease (SD) of ≥8 weeks
Durable clinical benefit (DCB) | approximately 6 months
  DCB, defined as DoCB ≥180 days. Patients who have best overall response of PD or those having clinical benefit but DoCB lasting <180 days will be considered as "non-DCB."
Disease control rate (DCR) | approximately 6 months
  DCR (i.e., CR+PR+SD at ≥8 weeks), as assessed by the Investigator using RECIST v1.1.
Time to response (TTR) | approximately 6 months
  TTR, defined as the time from the date of randomization (or date of registration for Part A patients) to the assessment date of the first instance of an overall response of CR or PR.
Exposure-response relationships for DKN-01 as data permit. | approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Sirard, Study Director — Leap Therapeutics, Inc.
Locations (40):
- United States (25):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - UCLA, Los Angeles, California
  - Florida Cancer Specialists & Research Institute (FCS), Cape Coral, Florida
  - Florida Cancer Specialists & Research Institute, Fleming Island, Florida
  - Florida Cancer Specialists & Research Institute, Gainesville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Florida Cancer Specialists & Research Institute, Wellington, Florida
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Oncology Hematology Associates - Springfield, Springfield, Missouri
  - Northwell Health, Lake Success, New York
  - New York University, New York, New York
  - Cornell University, New York, New York
  - Mount Sinai Medical Center - New York, New York, New York
  - White Plains Hospital, White Plains, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Tennessee Oncology, Chattanooga, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Germany (5):
  - Universitaetsklinikum Hamburg-Eppendorf (UKE) - Universitaeres Cancer Center Hamburg (UCCH), Hamburg
  - Universitaetsklinikum Heidelberg (UKHD) - Nationales Centrum fuer Tumorerkrankungen Heidelberg (NCT), Heidelberg
  - SLK-Kliniken Heilbronn GmbH - Klinikum am Gesundbrunnen - Klinik fuer Innere Medizin III, Heilbronn
  - Gemeinschaftspraxis fuer Haematologie und Onkologie - Magdeburg, Magdeburg
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
- South Korea (10):
  - Dong-A University Medical Center, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - CHA University - Bundang CHA General Hospital, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea - St. Vincent's Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No